CLINICAL TRIAL: NCT06867835
Title: A Phase 4, Open-Label Study of a Single Dose of Vyleesi® (Bremelanotide Injection) in Healthy, Premenopausal Lactating Female Subjects to Measure the Concentration of Bremelanotide in Breast Milk
Brief Title: Single Dose of Vyleesi in Lactating Female Subjects to Measure the Concentration of Bremelanotide in Breast Milk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cosette Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMR 3635-3
Record Dates: First submitted 2025-02-19; First posted 2025-03-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lactating Mother
MeSH Terms: interventions — bremelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vyleesi (Experimental): One dose of BMT 1.75 mg SC on Day 1
  Interventions: Drug: Vyleesi (Bremelanotide Injection)

INTERVENTIONS:
Drug: Vyleesi (Bremelanotide Injection) — Single dose of BMT 1.75 mg SC on Day 1

SUMMARY:
The primary objectives of this clinical trial performed with Vyleesi (Bremelanotide Injection) are:

* to evaluate if Bremelanotide (BMT) is secreted in breast milk of lactating women treated with a single dose of BMT 1.75 mg SC.
* to measure the concentration and characterize the pharmacokinetics of BMT secreted in breast milk of lactating women treated with a single dose of BMT 1.75 mg SC.

This open-label, pharmacokinetic (PK) study will be performed in 10 healthy lactating female subjects between 10 days and 6 months post-partum (inclusive). The maximum duration of subject participation in the study will be approximately 29 days, consisting of 3-week Screening period, a 1 day treatment period, and up to a 7 day follow-up period.

ELIGIBILITY:
Inclusion Criteria (Main Criteria):

* Female subjects ≥18 to 55 years of age (inclusive) and premenopausal
* Lactating, between 10 days and 6 months postpartum (inclusive).
* Exclusively breastfeeds their infant prior to participation in the study
* Is willing to pump and store breastmilk for feeding her infant for a minimum of 48 hours in advance of study initiation and discontinue breastfeeding their infant for the duration of their study participation (beginning from time of dosing with BMT) and a minimum of 24 hours following the Safety Follow-Up visit (i.e., a minimum of 48 hours following dosing with BMT).
* Ensure at the time of screening that the breastfed infant can feed from a bottle during maternal participation in the study
* The subject is not pregnant, and does not intend to become pregnant before, during, or within 1 complete menstrual cycle or 2 months after administration of study drug
* Subjects of childbearing potential who are sexually active with a nonsterilized male partner must have stable, continuous use of an acceptable method of contraception throughout the duration of the study, and for at least 60 days after the dose of study drug

Exclusion Criteria (Main Criteria):

* Breastfeeding is not well established in the mother-infant pair (e.g., poor latching of the infant or low milk supply).
* Any condition that interferes with the successful collection of milk from one or both breasts including but not limited to lactation mastitis (typically presents as a tender, hot, swollen area of the breast that may or may not involve an infection), milk blister that may present as a blocked nipple pore, breast abscess, etc.
* Has used any investigational compound and/or an experimental medical device within 28 days before Screening.
* Has taken BMT within 24 hours of participation in the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Lactating mother
Enrollment: 10 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Levels of Bremelanotide (BMT) in Breast Milk Over 24h After Administration of Vyleesi | 24 hours
  The levels/concentrations of bremelanotide (BMT) will be measured in breast milk samples collected at different timepoints up to 24h from lactating women who receive a single dose of Vyleesi (BMT 1.75 mg SC).
Area under the curve from time 0 to end of dosing interval (AUCtau) for BMT in Breast Milk | 24 hours
Maximum observed concentration (Cmax) of BMT in breast milk | 24 hours
Time to reach Cmax of BMT in breast milk (Tmax) | 24 hours
Terminal half-life of BMT in breast milk (t1/2) | 24 hours

SECONDARY OUTCOMES:
Levels of Bremelanotide (BMT) in Plasma Over 24h After Administration of Vyleesi | 24 hours
Area under the curve from time 0 to end of dosing interval (AUCtau) for BMT in Plasma | 24 hours
Maximum observed concentration (Cmax) of BMT in Plasma | 24 hours
Time to reach Cmax of BMT in Plasma (Tmax) | 24 hours
Milk:plasma ratio (M/P) of BMT Levels | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- First Excellence Research Group LLC, Doral, Florida, United States